CLINICAL TRIAL: NCT02022878
Title: Development of Computed Tomography Angiography Prediction Score for Percutaneous Revascularization of Chronic Total Occlusions: Multicenter CT-RECTOR Registry
Brief Title: Computed Tomography Angiography Prediction Score for Percutaneous Revascularization of Chronic Total Occlusions
Acronym: CT-RECTOR
Status: Completed | Type: Observational
Sponsor: Kerckhoff Heart Center (Other)
Collaborators: University of Giessen (Other); University Hospital Erlangen (Other); National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Principal Investigator, Prof. Dr. Christian W. Hamm, Director, Cardiology Department, Kerckhoff Heart Center
Other Study IDs: NP-0021-106/1416/13
Record Dates: First submitted 2013-12-22; First posted 2013-12-30 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Coronary Artery Disease
Keywords: Chronic total occlusion; Percutaneous coronary intervention; Coronary computed tomography angiography; Coronary angiography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Attempted PCI of CTO: Attempted PCI of CTO with preprocedural coronary CTA scan
  Interventions: Procedure: PCI of CTO

INTERVENTIONS:
Procedure: PCI of CTO

SUMMARY:
Chronic total occlusions (CTO) are encountered in almost one-fourth of patients undergoing coronary angiography. The presence of an untreated CTO has been related to adverse clinical prognosis, both in stable angina and acute myocardial infarction, and is often associated with persistent symptomatic angina. Depending on their symptomatic and functional status as well as anatomical complexity, CTO can be treated by optimal medical therapy only or therapy combined with coronary revascularization.

The potential benefits of percutaneous coronary intervention (PCI) in CTO include symptom relief, improved left ventricular function, and potentially a survival advantage associated with success when compared with failed revascularization. Of note, marked advances in endovascular techniques and device technology have resulted in substantial improvements of procedural success rates of PCI in CTO.

In spite of these advances, the vast majority of patients with CTO are still being managed medically or referred for coronary bypass surgery rather than PCI. The most common reason for deferring PCI in patients with CTO appears to be the uncertainty of predicting the procedural outcome of percutaneous revascularization. Further barriers to attempting CTO by PCI include the difficulty of gauging the time required for the procedure and the use of resources.

The CT-RECTOR (Computed Tomography REgistry of Chronic Total Occlusion Revascularization) study was designed to evaluate the application of coronary computed tomography angiography (CTA) for the prediction of procedural outcome of PCI in CTO in an international patient population. The main purpose of this multicenter registry is to develop a noninvasive CTA-based prediction tool (CT-RECTOR Score) for grading CTO suitability for PCI.

DETAILED DESCRIPTION:
Coronary CTA has recently emerged as a valuable noninvasive tool to provide guidance during percutaneous treatment of CTO. The main advantages of coronary CTA in characterization of CTO include the 3-dimensional visualization of occlusion trajectory and morphology as well as the exact evaluation of calcifications. Despite this, and although prior single-center studies suggested a potential utility of individual coronary CTA-based CTO characteristics for predicting PCI, there has been no compiled prediction model for grading CTO suitability for PCI in a large cohort of patients.

The CT-RECTOR registry is a retrospective, multicenter observational study of patients undergoing preprocedural coronary CTA before attempted PCI of CTO between 2007 and 2013. The study was designed to enroll 250 consecutive patients at 4 high-volume cluster sites in 2 European countries. CT-RECTOR sites were chosen on the basis of adequate coronary CTA volume and PCI proficiency to reflect the state-of-the-art, ''real-life'' management of patients with CTO.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for attempted PCI of CTO as part of their standard of care
* Performance of coronary CTA with 64-detector rows or greater within 6 weeks before attempted PCI of CTO
* Native vessel or bypass graft de novo or in-stent restenosis CTO
* Angiographically defined CTO with TIMI flow 0 and estimated duration over 3 months (the duration of the occlusion was determined based on either a history of sudden chest pain, a previous myocardial infarction in the same target vessel territory, or the time between the diagnosis made from coronary angiography and subsequent PCI)

Exclusion Criteria:

* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients at multiple international centers undergoing preprocedural coronary CTA before attempted PCI of CTO between 2007 and 2013.
Sampling Method: Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2013-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Successful guidewire crossing through CTO within 30 min | Intraprocedural
  Successful guidewire crossing through CTO within 30 min (defined as the time from initial insertion of the guidewire into the coronary lumen to the time it was successfully crossed through the lesion or was pulled out of the lumen because of unsuccessful guidewire crossing)

SECONDARY OUTCOMES:
Successful guidewire crossing through CTO and restoration of flow | Intraprocedural
  Successful guidewire crossing through CTO and restoration of flow (<50% residual stenosis and TIMI 2-3 flow)
Successful guidewire crossing through CTO with implantation of stent and restoration of flow | Intraprocedural
  Successful guidewire crossing through CTO with implantation of stent and restoration of flow (<50% residual stenosis and TIMI 2-3 flow) without severe coronary dissection or perforation

CONTACTS AND LOCATIONS:
Overall Officials: Christian W. Hamm, Prof. Dr., Principal Investigator — Kerckhoff Heart Center
Locations (4):
- Germany (3):
  - Kerckhoff Heart Center, Bad Nauheim
  - University Clinic Erlangen, Erlangen
  - University Clinic Giessen and Marburg, Giessen
- Institute of Cardiology, Warsaw, Poland

REFERENCES:
- [Derived] Opolski MP, Achenbach S, Schuhback A, Rolf A, Mollmann H, Nef H, Rixe J, Renker M, Witkowski A, Kepka C, Walther C, Schlundt C, Debski A, Jakubczyk M, Hamm CW. Coronary computed tomographic prediction rule for time-efficient guidewire crossing through chronic total occlusion: insights from the CT-RECTOR multicenter registry (Computed Tomography Registry of Chronic Total Occlusion Revascularization). JACC Cardiovasc Interv. 2015 Feb;8(2):257-267. doi: 10.1016/j.jcin.2014.07.031. PMID 25700748